CLINICAL TRIAL: NCT05251142
Title: Effects of Plyometric Training on Vertical Jump and Dynamic Stability in Volleyball Players With Chronic Knee Pain
Brief Title: Plyometric Training in Volleyball Players With Chronic Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0427
Record Dates: First submitted 2022-02-20; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Chronic Knee Pain
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric training (Experimental): Jumps in place. Standing jumps. Multiple hops and jumps. Box drills. Depth jumps.
  Interventions: Other: Plyometric training
- General exercises (Active Comparator): Dumbbell Squat, Dumbbell Alternating Bench Press, Straight Arm Pulldowns, Dumbbell Front Raises, Reverse Flyes, Overhead Tricep Extensions, Dumbbell Bicep Curls, Jackknife Crunches, Oblique Crunches, External Rotation
  Interventions: Other: General exercises

INTERVENTIONS:
Other: Plyometric training — Jumps in place. Some examples include multiple vertical jumps while reaching an overhead object, squat jump, pike jump, or tuck jump.
  * Standing jumps. Examples include the single leg jump, maximal vertical jump ,standing long jump or lateral long jump.
  * Multiple hops and jumps. Examples would include multiple long jumps or cone hops performed in succession, such as 5 hops in a row
  * Box drills. Examples of these drills include box jumps ,repeated box jumps, and single leg box jumps.
  * Depth jumps. Examples include stepping off the box and landing, stepping off the box and jumping vertically immediately after landing, or stepping off the box, landing, and sprinting.
  Arms: Plyometric training
Other: General exercises — Dumbbell Squat: 3 sets of 15 reps, Dumbbell Alternating Bench Press: 3 sets of 15 reps, Straight Arm Pulldowns: 3 sets of 15 reps, Dumbbell Front Raises: 3 sets of 15 reps, Reverse Flyes: 3 sets of 15 reps, Overhead Tricep Extensions: 3 sets of 15 reps, Dumbbell Bicep Curls: 3 sets of 15 reps, Jackknife Crunches: 3 sets of 20 reps, Oblique Crunches: 3 sets of 20 reps, External Rotation: 3 sets of 15 reps
  Arms: General exercises

SUMMARY:
The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah Internatinal University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through random number generator by Non-probability Convenient random sampling technique. Subjects in Group A will receive plyometric training. Group B will receive general training.

DETAILED DESCRIPTION:
The objective of the study is to determine the effects of plyometric training on vertical jumps and dynamic stability in volleyball players with chronic knee pain.

The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah Internatinal University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through random number generator by Non-probability Convenient random sampling technique. Subjects in Group A will receive plyometric training. Group B will receive general training.

The outcome measures will be assessed by Vertical jump test, Hop test and Y balance test

The data will be analyzed by SPSS, version 25. Statistical significance is P= 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Both genders. Age between 15 to 30 years ACR criteria for knee OA. BMI less than 30

Exclusion Criteria:

* Players with open wounds. Players with diabetes. Grade IV OA on kellergan Lawrence. Any traumatic condition that can hinder polymetric training. Ankle instability sprain/ strain.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-10 (Estimated)

PRIMARY OUTCOMES:
Vertical Jump Test | 4 weeks
  The Vertical Jump test is designed to measure an athlete's lower body strength
Hop Test | 4 weeks
  In this test, the aim is to jump as far as possible on a single leg, without losing balance and landing firmly.
Y Balance Test | 4 weeks
  This is a portion of the Functional Movement Systems screen used to evaluate dynamic balance and functional symmetry in order to determine a person's risk for injury or return to sport readiness.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Atif Javed, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- D.G. Khan Sports Complex, Dera Ghazi Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alikhani R, Shahrjerdi S, Golpaigany M, Kazemi M. The effect of a six-week plyometric training on dynamic balance and knee proprioception in female badminton players. J Can Chiropr Assoc. 2019 Dec;63(3):144-153. PMID 31988535
- [Background] Shams F, Hadadnezhad M, Letafatkar A, Hogg J. Valgus Control Feedback and Taping Improves the Effects of Plyometric Exercises in Women With Dynamic Knee Valgus. Sports Health. 2022 Sep-Oct;14(5):747-757. doi: 10.1177/19417381211049805. Epub 2021 Oct 15. PMID 34651505
- [Background] Lee HM, Oh S, Kwon JW. Effect of Plyometric versus Ankle Stability Exercises on Lower Limb Biomechanics in Taekwondo Demonstration Athletes with Functional Ankle Instability. Int J Environ Res Public Health. 2020 May 22;17(10):3665. doi: 10.3390/ijerph17103665. PMID 32456048
- [Background] Hammami M, Ramirez-Campillo R, Gaamouri N, Aloui G, Shephard RJ, Chelly MS. Effects of a Combined Upper- and Lower-Limb Plyometric Training Program on High-Intensity Actions in Female U14 Handball Players. Pediatr Exerc Sci. 2019 Nov 1;31(4):465-472. doi: 10.1123/pes.2018-0278. Epub 2019 Jul 17. PMID 31310989
- [Background] Al Attar WSA, Husain MA. The effect of combining plyometrics exercises and balance exercises in improving dynamic balance among female college athletes: A randomized controlled trial. PM R. 2022 Oct;14(10):1177-1187. doi: 10.1002/pmrj.12690. Epub 2021 Sep 14. PMID 34375501
- [Background] Zhao W, Wang C, Bi Y, Chen L. Effect of Integrative Neuromuscular Training for Injury Prevention and Sports Performance of Female Badminton Players. Biomed Res Int. 2021 Apr 23;2021:5555853. doi: 10.1155/2021/5555853. eCollection 2021. PMID 33987438